CLINICAL TRIAL: NCT06287762
Title: A Single-Center Prospective Natural History Study of RYR1-Related Disorders
Brief Title: A Natural History Study of RYR1-Related Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10001737; 001737-CC
Record Dates: First submitted 2024-02-29; First posted 2024-03-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Ryanodine Receptor 1-Related Myopathy; Ryanodine Receptor 1 Related Disorders
Keywords: RYR1; Muscle Disease; Natural History; Congenital Myopathy
MeSH Terms: conditions — Muscular Diseases; Myotonia Congenita

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Centralized: Visits are conducted at the NIH clinical center. All participants are ambulatory.
- Decentralized: Visits are conducted via telehealth.

SUMMARY:
Background:

Congenital myopathies (CM) are genetic disorders that can cause decreased muscle tone and muscle weakness. Most CMs in the United States are related to the ryanodine receptor 1 (RYR1) gene. Researchers need more natural history data to learn about these CMs in children and adults.

Objective:

To learn more about the signs, symptoms, and course of RYR1-related disorders.

Eligibility:

People aged 7 years and older with an RYR1-related disorder.

Design:

Ambulatory participants will come to the Clinical Center and non-ambulatory participants will visit via telehealth.

Visits will be once a year for 3 or 5 years. Clinical Center visits will take 2 to 3 days.

All participants will undergo tests including:

Photos and videos. These will be taken to document the participant s condition.

Blood and urine tests.

Activity Tracker. Participants will wear a device to record their activity.

Questionnaires. Participants will answer questions about their health, pain, fatigue, stress, quality of life, and other topics.

Participants who visit the Clinical Center will also undergo:

Tests of heart and lung function.

Motor skills and strength tests. Participants will walk, climb stairs, kneel, crawl, stand up, and perform other movements to test their strength and abilities. They will squeeze and pinch a handheld device to test their grip.

Imaging scans.

Skin biopsy. Adult participants may opt to have a sample of skin taken (one time only).

Eye exam

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

This prospective natural history study seeks to characterize the clinical manifestations and course of Ryanodine Receptor 1 -related disorders (RYR1-RD). RYR1-RD include a wide range of rare congenital and adult-onset neuromuscular phenotypes that are typically slowly progressive. The study is observational and comprises a primary data collection phase (Years 1-3) and extended follow-up phase (Years 4-5), stratified into centralized (ambulatory) and decentralized (non-ambulatory) arms. During each phase, there will be one visit per year. The study will enhance the foundational knowledge of RYR1-RD and support clinical trial readiness.

OBJECTIVE:

Primary:

Characterize phenotype and disease course over a three-year period

Secondary:

Characterize phenotype and disease course over an extended (2-year) period (total 5 years)

Exploratory:

1. Investigate potential biomarkers of disease status and progression
2. Explore clinical meaningfulness thresholds for research assessments
3. Extract common data elements from existing medical records (real-world evidence)

   ENDPOINTS:

   Primary:

   Change from baseline to Year 3 in:

   Motor function and performance
   * Motor Function Measure (MFM) sub-domains (percent of maximum score)
   * Six-minute walk test (meters travelled with percent predicted)
   * Timed functional tests (ascend four stairs, descend four stairs, supine to stand) (seconds)
   * Grip and pinch strength (kg and percent predicted)
   * Performance of Upper Limb (PUL)
   * Accelerometry (wearable sensor)
   * Quantitative muscle assessment
   * Brooke and Vignos assessment

   Pulmonary function
   * Forced vital capacity (percent reference norm)
   * Forced expiratory volume at 1 second (percent reference norm)
   * Slow vital capacity (Liters)
   * Maximal voluntary ventilation (Liters)
   * Maximum inspiratory pressure (MIP)
   * Maximum expiratory pressure (MEP)

   Patient-reported outcomes
   * PROMIS-57 Profile (subscale and overall t-scores); adults - depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and satisfaction with participation in social roles
   * PROMIS Ped-25 Profile (subscale and overall t-scores); 8 - 17 y
   * PROMIS Parent Proxy 25 Profile - Fatigue, physical stress experiences, positive affect and wellbeing, psychological stress experiences, anxiety/fear, physical function, pain; 5 - 7 y
   * PROMIS Upper Extremity - Short Form 7a
   * PROMIS Pediatric Upper Extremity - Short Form 8a
   * PROMIS Parent Proxy Upper Extremity - Short Form 8a
   * Physical Activity Questionnaire for Children (PAQ-C); 8 - 13 y
   * Physical Activity Questionnaire for Adolescents (PAQ-A); 14 - 17 y
   * International physical activity questionnaire (IPAQ); adults

   Ophthalmology
   * Visual acuity
   * Dilated ophthalmology exam at baseline only
   * Extraocular motility assessment
   * Marginal reflex distance (Ptosis)
   * Optical Coherence Tomography
   * Ancillary testing, imaging, and repeat dilated exams as indicated, based on assessment and discretion of clinician

   Secondary:

   Change from baseline to Year 5 in:

   Motor function and performance
   * Motor Function Measure (MFM) sub-domains (percent of maximum score)
   * Six-minute walk test (meters travelled with percent predicted)
   * Timed functional tests (ascend four stairs, descend four stairs, supine to stand) (seconds)
   * Grip and pinch strength (kg and percent predicted)
   * Performance of Upper Limb (PUL)
   * Accelerometry (wearable sensor)
   * Quantitative muscle assessment
   * Brooke and Vignos assessment

   Pulmonary function
   * Forced vital capacity (percent reference norm)
   * Forced expiratory volume at 1 second (percent reference norm)
   * Slow vital capacity (Liters)
   * Maximal voluntary ventilation (Liters)
   * Maximum inspiratory pressure (MIP)
   * Maximum expiratory pressure (MEP)

   Patient-reported outcomes
   * PROMIS-57 Profile (subscale and overall t-scores); adults - depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and satisfaction with participation in social roles
   * PROMIS Ped-25 Profile (subscale and overall t-scores); 8 - 17 y
   * PROMIS Parent Proxy -25 Profile Fatigue, physical stress experiences, positive affect and wellbeing, psychological stress experiences, anxiety/fear, physical function, pain; 5 - 7 y
   * PROMIS Upper Extremity - Short Form 7a
   * PROMIS Pediatric Upper Extremity - Short Form 8a
   * PROMIS Parent Proxy Upper Extremity - Short Form 8a
   * Physical Activity Questionnaire for Children (PAQ-C); 8 - 13 y
   * Physical Activity Questionnaire for Adolescents (PAQ-A); 14 - 17 y
   * International physical activity questionnaire (IPAQ); adults

   Ophthalmology
   * Visual acuity
   * Dilated ophthalmology exam at baseline only
   * Extraocular motility assessment
   * Marginal reflex distance (Ptosis)
   * Optical Coherence Tomography
   * Ancillary testing, imaging, and repeat dilated exams as indicated, based on assessment and discretion of clinician

   Exploratory:

   Biomarkers

   Including but not limited to:
   * Plasma NAD plus, NADH
   * Plasma GSH, GSSG
   * Plasma cytokines
   * Serum creatine phosphokinase
   * Urine and plasma 15-F2t isoprostane
   * Urine 8OHdG
   * PBMC (Peripheral Blood Mononuclear Cell)
   * Near infrared spectroscopy (muscle tissue oxygenation)
   * Dixon MRI of lower extremity
   * Optional skin punch biopsy (fibroblast culture)
   * Muscle ultrasound
   * Electrical impedance myography (EIM)

ELIGIBILITY:
* INCLUSION CRITERIA (CENTRALIZED ARM)

  1. Stated willingness to comply with all study procedures, availability for the duration of the study, and submission of medical records to research team prior to screening.
  2. Male or female, aged >=7 years of age.
  3. Genetically confirmed RYR1-related disorder, evidenced by pathogenic or likely pathogenic variants identified by CLIA testing (whole genome, exome, targeted, partial or full RYR1 sequencing) OR variant of uncertain significance with supporting clinical phenotype.
  4. Agreement to adhere to Lifestyle Considerations throughout study duration.
  5. Ability of subject to communicate their understanding of the purpose of the study, and willingness to provide assent and/or to sign a written informed consent document.
  6. Resides in the United States.

EXCLUSION CRITERIA (CENTRALIZED ARM)

1. Participation in an IND, IDE, or equivalent clinical study in the past six months
2. Severe disability or mobility issues (inability to walk 10 meters with or without assistance)
3. Requires mechanical ventilation or tracheotomy
4. Other neuromuscular diseases resulting in muscle weakness
5. Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study (e.g. active infection) or safety of the subject.

INCLUSION CRITERIA (DE-CENTRALIZED ARM)

1. Stated willingness to comply with all study procedures, availability for the duration of the study, and submission of medical records to research team prior to screening.
2. Male or female, aged > 7 years of age.
3. Genetically confirmed RYR1-related disorder, evidenced by pathogenic or likely pathogenic variants identified by CLIA testing (whole genome, exome, targeted, partial or full RYR1 sequencing) OR variant of uncertain significance with supporting clinical phenotype.
4. Ability of subject to communicate their understanding of the purpose of the study, and willingness to provide assent and/or sign a written informed consent document.
5. Resides in the United States

EXCLUSION CRITERIA (DE-CENTRALIZED ARM)

1. Participation in an IND, IDE, or equivalent clinical study in the past six months
2. Other neuromuscular diseases resulting in muscle weakness
3. Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study (e.g. active infection) or safety of the subject

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 150 clinically stable adults and children (7 years of age or older) with genetically confirmed RYR1-RD.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse and disease-related events | 3 years
  Serious (21CFR312.32) adverse events:- Narrative description (clinician)- Causality assessment (related or unrelated to disease)- CTCAE system organ class- CTCAE lower-level term- Falls questionnaire; adults
Medical data review | 3 years
  - Demographics- Developmental history- Medical history- Social determinants of health (environmental conditions such as economic stability, health care and education access and quality, neighborhood and built environment, and social and community context.- Full physical exam- Review of genetic diagnostic report/results- Prior medical records
Ophthalmology | 3 years
  - Marginal reflex distance (Ptosis)- Binocular horizontal visual field test- Optical Coherence Tomography- Goldmann Perimetry Degrees: lateral rectus, superior rectus, inferior oblique, medial rectus, superior oblique, inferior rectus
Patient-reported outcomes | 3 years
  - PROMIS-57 Profile (subscale and overall t-scores); adults - depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and satisfaction with participation in social roles- PROMIS Ped-25 Profile (subscale and overall t-scores); 8 - 17 y- PROMIS Parent Proxy 25 Profile - Fatigue, physical stress experiences, positive affect and wellbeing, psychological stress experiences, anxiety/fear, physical function, pain; 5 - 7 y- PROMIS Upper Extremity - Short Form 7a- PROMIS Pediatric Upper Extremity - Short Form 8a- PROMIS Parent Proxy Upper Extremity - Short Form 8a- Physical Activity Questionnaire for Children (PAQ-C); 8 - 13 y- Physical Activity Questionnaire for Adolescents (PAQ-A); 14 - 17 y- International physical activity questionnaire (IPAQ); adults
Pulmonary function | 3 years
  - Forced vital capacity (% reference norm)- Forced expiratory volume at 1 second (% reference norm) - Slow vital capacity (Liters)- Maximal voluntary ventilation (Liters)- Maximum inspiratory pressure (MIP)- Maximum expiratory pressure (MEP)
Motor function and performance | 3 years
  - Motor Function Measure (MFM) sub-domains (percent of maximum score)- Six-minute walk test (meters travelled with percent predicted)- Timed functional tests (ascend four stairs, descend four stairs, supine to stand) (seconds)- Grip and pinch strength (kg and percent predicted)- Performance of Upper Limb (PUL)- Accelerometry (wearable sensor)- Quantitative muscle assessment- Brooke and Vignos assessment

SECONDARY OUTCOMES:
Characterize phenotype and disease course over an extended (2-year) period (total 5 years).Collect exploratory biomarker data. | 5 years
  (1) Investigate potential biomarkers of disease status and progression(2) Explore clinical meaningfulness thresholds for research assessments(3) Extract common data elements from existing medical records (real-world evidence)

CONTACTS AND LOCATIONS:
Overall Officials: Tokunbor A Lawal, C.R.N.P., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001737-CC.html